CLINICAL TRIAL: NCT04516525
Title: Assessment of the Impact of Resynchronization Therapy on Renal Function
Brief Title: The Impact of CRT on Renal Function
Status: Completed | Type: Observational
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Agnieszka Gala-Bladzinska, Principal Investigator, University of Rzeszow
Other Study IDs: 1/AGB
Record Dates: First submitted 2020-08-06; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Chronic Kidney Diseases; Chronic Heart Failure
Keywords: Chronic cardio-renal syndrome biomarkers
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples Without DNA — blood, urina
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: cardiac resynchronisation therapy (CRT) implantation — In a group of 100 patients with chronic cardio-renal syndrome, the blood and urine biomarkers are tested before CRT implantation and after 48 hours, 3 months and 1 year of follow-up.

SUMMARY:
The study is observational, prospective, including patients undergoing CRT-D / CRT-P implantation in the department of cardiology. In the current project, the researchers assumed that the improvement in cardiac function obtained in patients qualified according to the ESC / PTK guidelines for resynchronization therapy may improve renal function in a prospective 12-month follow-up. In addition, it is planned to take into account the possibility of temporary deterioration of kidney function, which may occur immediately after implantation of the resynchronization device due to the nephrotoxic effect of the contrast agent.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with heart failure who had met the criteria for CRT implantation according to European Society of Cardiology guidelines for the treatment of heart failure

Exclusion Criteria:

* no written consent to participate in the study
* no indications for CR implantation
* current infection
* children
* pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with heart failure who had met the criteria for CRT implantation according to European Society of Cardiology guidelines for the treatment of heart failure
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of changes renal function: 48 hours, one month and one year after cardiac resynchronization therapy device implantation procedure. | 1 year for each patient in the study
  Assessment of the number of patients with with chronic type 2 cardio-renal syndrome with improvement or deterioration renal function assessed by blood and urine biomarkers within the first 48 hours, one month and one year after CRT implantation.

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed in the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Gala-Bladzinska A, Romanek J, Mazur D, Stepek T, Braun M, Szafarz P, Chlebus M, Przybylski A. Reduced Albuminuria and Potassemia Indicate Early Renal Repair Processes after Resynchronization Therapy in Cardiorenal Syndrome Type 2. Cardiol Res Pract. 2020 Mar 21;2020:2727108. doi: 10.1155/2020/2727108. eCollection 2020. PMID 32274209